CLINICAL TRIAL: NCT01710592
Title: A Randomised Phase II Trial of Epirubicin, Oxaliplatin and Capecitabine (EOX) Versus Docetaxel and Oxaliplatin (ElTax) in the Treatment of Advanced Gastro-oesophageal Cancer
Brief Title: A Phase II Trial of Epirubicin, Oxaliplatin and Capecitabine (EOX) Versus Docetaxel and Oxaliplatin (ElTax) in the Treatment of Advanced Gastro-oesophageal Cancer
Acronym: ELECT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICORG 06-05; NCT00806949 (obsolete NCT alias)
Record Dates: First submitted 2012-10-15; First posted 2012-10-19 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Gastro Oesophageal Cancer
MeSH Terms: interventions — Epirubicin; Oxaliplatin; Capecitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epirubicin, Oxaliplatin, Capecitabine (Active Comparator): * Epirubicin 50mg/m2 (day 1) bolus injection
  * Oxaliplatin 130mg/m2 (day 1) in 250mls of 5% dextrose. i.v. over 2 hours
  * Capecitabine 625mg/m2 (days 1-21) b.d. orally
  * 8 x 3-weekly cycle
  Interventions: Drug: Epirubicin; Drug: Oxaliplatin; Drug: Capecitabine
- Docetaxel, Oxaliplatin (Active Comparator): * Docetaxel 20mg/m2 (days 1, 8 & 15)in 250mls of 5% dextrose. i.v. over 30mins (Dexamethasone 8mg i.v, Chlorpheniramine 10mg i.v,Ranitidine 50mg i.v. to be given 30 minutes prior to Docetaxel)
  * Oxaliplatin 85mg/m2 (days 1 & 15)in 250mls of 5% dextrose. i.v. over 2 hours
  * 6 x 4-weekly cycle
  Interventions: Drug: Oxaliplatin; Drug: Docetaxel

INTERVENTIONS:
Drug: Epirubicin
  Arms: Epirubicin, Oxaliplatin, Capecitabine
Drug: Oxaliplatin
Drug: Capecitabine
  Arms: Epirubicin, Oxaliplatin, Capecitabine
Drug: Docetaxel
  Arms: Docetaxel, Oxaliplatin

SUMMARY:
Whilst oxaliplatin and docetaxel have established activity in the treatment of advanced gastro-oesophageal cancer, their role, however, in the management of this disease remains unclear. Furthermore it is unclear whether this disease is optimally treated with a combination of two or three cytotoxic drugs. This trial aims to determine whether the combination of oxaliplatin and weekly docetaxel warrants further investigation in a formal phase III trial. The combination of epirubicin, oxaliplatin and capecitabine will be the comparator arm for this evaluation.

Primary Objective:

Determine in a randomised study if the response rate to docetaxel and oxaliplatin (ElTax) is comparable to epirubicin, oxaliplatin and capecitabine (EOX) and warrants further evaluation in advanced gastro-oesophageal cancer.

Secondary Objective:

To examine the effect of treatment on time to progression, progression free survival, overall survival, quality of life, and the associated toxicity from treatment.

DETAILED DESCRIPTION:
This is a randomised two-arm parallel group phase II study. 140 patients will be recruited over a period of 12 months, and will be randomised to receive either eight 3-weekly cycles of Epirubicin, Oxaliplatin and Capecitabine (EOX) or six 4-weekly cycles of Docetaxel and Oxaliplatin (EITax).

ELIGIBILITY:
Inclusion Criteria:

* Unresectable or metastatic, histologically confirmed adenocarcinoma of the stomach, gastro-oesophageal junction or lower third of the oesophagus with measurable disease on CT scanning (see RECIST Criteria, Appendix C of the protocol for definition of measureable disease).
* No previous treatment for advanced disease (previous adjuvant/neo-adjuvant treatment acceptable if >12 months previously).
* Absence of serious concomitant illness (i.e. MI within previous 6 months), uncontrolled angina, uncontrolled hypertension, severe COPD (>3 admissions for infective exacerbation in past 12 months) etc.
* ECOG performance status ≤ 2.
* Age ≥ to 18.
* Life expectancy ≥ 3 months
* Adequate renal, hepatic and bone marrow function
* Creatinine clearance ≥ 50 ml/min as calculated using the Cockcroft and Gault formula (see Appendix L).
* Liver function tests:

Bilirubin ≤ 1.0 x ULN, AST ≤ 1.5 x ULN, ALT ≤ 1.5 x ULN,Haemoglobin > 10.0 g/dl, Absolute neutrophil count >1.5 x 109 /L, Platelet count > 100 x109/L.

•Before randomisation, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Symptoms or signs of peripheral neuropathy.
* Patients known to have second or third degree heart block.
* Previous or concurrent malignancy, with the exception of basal cell carcinoma of the skin or in-situ neoplasia of the uterine cervix.
* Known hypersensitivity to taxanes, oxaliplatin, or fluoropyrimidines.
* Pregnant or nursing.
* Female of child-bearing potential, or male partner of female of child bearing potential not taking adequate contraceptive precautions.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-05; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Determine in a randomised study if the response rate to docetaxel and oxaliplatin (ElTax) is comparable to epirubicin, oxaliplatin and capecitabine (EOX) and warrants further evaluation in advanced gastro-oesophageal cancer | Two Years

SECONDARY OUTCOMES:
In addition we will examine the effect of treatment on time to progression. | Two Years
To examine the associated toxicity from treatment | 2 years
To examine the effect of treatment on survival | 2 years
To examine the effect of treatment on Quality of life. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Eatock, Dr, Principal Investigator — Cancer Trials Ireland
Locations (6):
- Ireland (6):
  - Mercy University Hospital, Cork
  - Beaumont Hospital, Dublin
  - Mater Misericordiae University hospital & Mater Private Hospital, Dublin
  - St James's Hospital, Dublin
  - The Adelaide and Meath Hospital, Dublin
  - Waterford Regional Hospital, Waterford